CLINICAL TRIAL: NCT06217718
Title: The Effect of Empowerment Model-Based Telenursing Interventions in Empowering Patients With COPD
Brief Title: The Effect of Telenursing Interventions in Empowering Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahide Aksoy (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Zahide Aksoy, Lecturer, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MarmaraU-HEM-ZA-01
Record Dates: First submitted 2024-01-07; First posted 2024-01-22 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Copd; Empowerment; Empowerment, Patient; Self Efficacy
Keywords: telenursing; empowerment; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Empowerment; Patient Participation

STUDY DESIGN:
Intervention Model Description: Two groups with experimental and control groups
Who Masked: Participant, Outcomes Assessor
Masking Description: In order to prevent selection bias in the study, the assignment to the experimental and control groups will be made on a computer by a person who is unfamiliar with the research process. Individuals included in the study will not be told whether they are in the experimental or control group. The analysis of the data will be done by a statistics expert who is outside the research process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telenursing Interventions Group (Experimental): Participants in this group will receive five hours of face-to-face empowerment training. After the training, the experimental group will be monitored remotely by the researcher nurse via tele-nursing interventions for 12 weeks. Participants will be given a pulse oximeter, symptom diary, action plan, oxygen saturation-pulse monitoring chart. Participants will be asked to measure their oxygen saturation and pulse once a day for 12 weeks and record it on the chart. Participants will also be asked to record their complaints in their symptom diary. Participants will be called by the researcher every two weeks (on Thursdays) and informative and reminding text messages prepared specifically for the disease will be sent to the participants three times a week for 12 weeks. Participants will be able to reach the researchers by phone whenever they need.
  Interventions: Other: Telenursing Interventions
- No Intervention Group (No Intervention): Participants in this group will be given a pulse oximeter, symptom diary, action plan, oxygen saturation-pulse monitoring chart. No intervention will be taken.

INTERVENTIONS:
Other: Telenursing Interventions — Patient follow-up with phone calls and text messages
  Arms: Telenursing Interventions Group

SUMMARY:
The aim of this study is to evaluate the effect of telenursing interventions based on the empowerment model in empowering patients with COPD.

DETAILED DESCRIPTION:
Patient empowerment is gaining importance and popularity day by day as it can be sustained through telehealth applications. The importance of using communication technologies in providing health care services has become more evident during the COVID-19 pandemic. When integrated into healthcare, technology-centric services provide continuous and easily accessible health data for patients and help facilitate self-monitoring. With tele-nursing, COPD patients can be strengthened in health literacy by teaching them how to access accurate and reliable resources. Through tele-nursing, online support groups and forums can be created among COPD patients so that patients can share their experiences with each other. In this way, social support is provided to patients who have to remain in social isolation due to their illness.

ELIGIBILITY:
Inclusion Criteria:

* Having a confirmed COPD diagnosis for at least one year
* being literate,
* Having the cognitive and mental competence to answer questions,
* Being able to use a mobile phone,
* Disease symptoms are at a level that does not interfere with communication,
* Being in COPD Stage 2 and Stage 3 according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD: Global Initiative for Chronic Obstructive Lung Disease) criteria (30% ≤ FEV1 <80% (of expected)),

Exclusion Criteria:

* The disease is in the acute exacerbation period,
* Dyspnea is at a level that prevents cooperation,
* Having sensory loss regarding vision, hearing and speech,
* Refusal to sign informed consent forms
* It is the refusal of the research to complete the data collection tools.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
COPD Empowerment Scale | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  A 31-item scale that evaluates the impact of interventions on individuals with COPD.

SECONDARY OUTCOMES:
Lung Function Test | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  A spirometri test that evaluates lung capacity. FEV1 values will increase after the intervention.
COPD Assesment Test | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  It is an eight-item test that measures the effects of COPD and deterioration in health status. CAT assessment test score; 0-10 is low 11-20 is considered medium effective, 21-30 is considered highly effective, and 31-40 is considered very high effective.
Number of hospital admissions due to COPD exacerbation | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  The number of hospital admissions due to COPD exacerbation in the experimental group will decrease.
Number of hospitalizations due to COPD exacerbation | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  The number of hospitalizations due to COPD exacerbation in the experimental group will decrease.
Modified Barthel Index | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  A scale that evaluates physical competence and independence in daily living activities. It evaluates 0-15 points with 10 items. On this scale, where the possible score varies between 0 and 100, the higher the score, the more independent the patient is from other people.
Modified Medical Research Council | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  A brief 5-item scale describing dyspnea. Scores between 0 and 1 are considered mild, and scores of 2 and above are considered moderate to severe dyspnea.
Inhaler Device Use Skill Scale | Pre-test, Post-test (3rd month), Follow-up Test (6th month)
  An observational test that measures inhaler device usage skill, with 10 usage steps explained. 1 point for correct use of each item; Incomplete or incorrect use is given 0 points.

CONTACTS AND LOCATIONS:
Overall Officials: Zahide Aksoy, MSc, Principal Investigator — Marmara University; Saime Erol, Ph.D, Study Director — Marmara University; Özlem Oruç, M.D, Study Director — Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital
Locations (1):
- Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aksoy Z, Erol S, Oruc O. Effects of empowerment model-based telenursing interventions on empowerment in individuals with COPD. BMC Nurs. 2025 Dec 19;25(1):52. doi: 10.1186/s12912-025-04225-z. PMID 41420230